CLINICAL TRIAL: NCT03364881
Title: Multicenter Clinical Trial of Anatomical Classifications of Henle's Trunk in Laparoscopic Right Hemi-colectomy.
Brief Title: Anatomical Classifications of Henle's Trunk
Acronym: HeLaRC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Sponsor
Other Study IDs: ShanghaiMISC
Record Dates: First submitted 2017-12-01; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-11

CONDITIONS: Mesenteric Vein; Colorectal Surgery; Henle's Trunk

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Right colon has complicated anatomy which is surrounded by important organs. The variations of vessels are more frequent than in left colon, which contribute to the difficulty of surgery. Among the variations, Henle's trunk is more obvious that makes it the commonest cause of bleeding during operation. Several veins can be found to conjoin the Henle's trunk, among which ASPDV and REGV are the two common tributaries while RCV,MCV,SRCV may vary from people to people. As a result, a better understanding of the anatomical classification of Henle's trunk is a must during operation. However, existing studies of Henle's trunk are very rare and often single-centered with minimal samples.In order to achieve better surgical outcome and reduce operative complications, the investigators design this study to investigate the anatomical classification of Henle's trunk and the surgical outcome of each type.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who undergoing laparoscopic right hemi-colectomy with D3 lymphadenectomy
2. Pathology: adenocarcinoma or high-grade intraepithelial neoplasia proven by colonoscopic biopsy.
3. Localization: tumor located between cecum and proximal 1/3 portion of transverse colon.
4. Patients have to be aware of the aim of the trial, and have signed the informed consent.

Exclusion Criteria:

1. History of any gastrointestinal surgery.
2. Patients with ileus, perforation, bleeding and any other conditions required of emergent surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is a prospective study，and based on the number of branches, the anticipant populations of this study is 500.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-11-17 (Actual); Primary Completion 2019-05-17 (Estimated); Study Completion 2020-05-17 (Estimated)

PRIMARY OUTCOMES:
classifications of Henle's trunk | 2 yeas
  based on the number of colic veins that conjoin the SMV

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ruijin Hospttal, Shanghai, Sahgnhai, China